CLINICAL TRIAL: NCT06602271
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of PF614 for the Treatment of Moderate to Severe Pain After Abdominoplasty
Brief Title: PF614 Analgesic Activity in Acute Postoperative Pain (PF614-301)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ensysce Biosciences (Industry)
Collaborators: Rho, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PF614-301
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain, Acute
Keywords: PF614, oxycodone, prodrug
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Pain intensity (11-point NRS) assessments at rest (NRS-R; minimum 3-minute rest) and with movement (NRS-A, where movement is defined as moving from a supine to sitting position) will be recorded at scheduled times during the inpatient period after Time 0 and immediately before each use of rescue medication.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PF614 25 mg (Experimental): Oral administration every 12 hours
  Interventions: Drug: PF614 capsule
- PF614 37.5 mg (Experimental): Oral administration every 12 hours
  Interventions: Drug: PF614 capsule
- PF614 50 mg (Experimental): Oral administration every 12 hours
  Interventions: Drug: PF614 capsule
- Placebo (Placebo Comparator): Oral administration every 12 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF614 capsule — Experimental oxycodone prodrug
  Arms: PF614 25 mg; PF614 37.5 mg; PF614 50 mg
Drug: Placebo — Inactive medication
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the analgesic activity of PF614 (an oral oxycodone prodrug extended-release analgesic) for control of postsurgical pain in subjects scheduled for abdominoplasty surgery. The main question to be answered is:

• To assess the analgesic efficacy of PF614 compared to placebo in subjects with moderate to severe pain following abdominoplasty.

Participants will be asked to take oral blinded doses of study medication at about one hour before surgery starts, and then every 12 hours after surgery for up to 4 days.

Participants will be asked to:

* Rate their pain on a 0-10 numerical rating scale (NRS) at various timepoints up to 5 days following surgery;
* Tell us about the need for rescue medication if they continue to have moderate-to-severe pain;
* Tell us about any side effects or adverse effects that they may experience to help us understand the safety and tolerability of the test medications;
* Provide periodic blood samples to help us understand how much study drug is in their system.

Participants will stay in a clinic setting and be monitored for safety for 5 days following surgery. We anticipate that participants will be discharged on Day 5, pending medical review, and then keep a diary to record study-related pain and adverse effects for an additional 2-4 days after discharge.

DETAILED DESCRIPTION:
This will be a Phase 3, multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of PF614 in the treatment of moderate to severe acute postoperative pain following abdominoplasty. The study will be conducted in 4 phases: Screening, Treatment, Outpatient and Follow-up.

Screening Phase Prospective participants will complete a standard medical screening within 28 days of the abdominoplasty procedure. At Screening, participants will provide written informed consent to participate in the study before any protocol-specified procedures or assessments are conducted.

Treatment Phase The Treatment Phase will begin on the day of the abdominoplasty procedure (Day 1) and will end on postoperative Day 5. Participants will be admitted to the study center on the morning of the scheduled procedure and will be confined throughout the Treatment Phase (5 days, 4 nights).

Days 1-4 (0-72 hours): Randomized Treatment Period Following admission to the study center, presurgical procedures will include participant training on pain intensity assessments, which will be administered as 11-point numerical rating scales (NRS). Participants who continue to meet all study entry criteria will be randomized prior to the abdominoplasty procedure in a 1:1:1:1 ratio to 1 of 4 treatment groups.

Treatment groups will include the following doses: PF614 25 mg, PF614 37.5 mg, PF614 50 mg, and Placebo.

The first dose of study drug will be administered 1 hour (±15 minutes) prior to the scheduled start time of the abdominoplasty procedure (i.e., prior to time of anesthetic induction). Time 0 is defined as the time of first study drug administration. Additional doses of study drug will be provided every 12 hours (BID) (±15 minutes), with the last scheduled study drug administration at 72 hours. Qualified medical personnel and/or investigators who are ACLS (Advanced Cardiovascular Life Support) certified will be present in the clinic during the inpatient treatment phase when participants are administered opioid medications.

Participants will undergo a full abdominoplasty procedure without liposuction or other collateral procedures under a standardized anesthetic protocol. Prior to wound closure, the surgeon will perform a transversalis abdominal plane (TAP) block by infiltrating 1% lidocaine with epinephrine 7 mg/kg with a maximum dose of 500 mg. Participants may be administered supplemental oxygen for at least the first 2 hours postoperatively (end of surgery defined as time of extubation), and the participant will be weaned as clinically appropriate.

Participants may receive hydrocodone/acetaminophen APAP (HC/APAP) 5 mg/325 mg every 6 hours as rescue medication, up to a maximum of 20 mg/1300 mg every 24 hours. If HC/APAP is administered, participants will not be eligible to receive additional HC/APAP for the following 6 hours.

Pain intensity (11-point NRS) assessments at rest (NRS-R; minimum 3-minute rest) and then with movement (NRS-A, where movement is defined as moving from a semi-supine or supine to sitting position without assistance) will be recorded at scheduled times (if participants are asleep, they will be awoken for scheduled assessments) during the inpatient period, and NRS-R and NRS-A will be recorded immediately before each use of rescue medication. Study drug will be administered after assessment of pain at each time point when dosing and pain assessments overlap. Pain intensity will also be recorded before early study discontinuation. Blood will be collected for pharmacokinetic (PK) analysis; observer-rated assessments of sedation (using the Modified Observer's Assessment of Alertness/Sedation Scale [MOAA/S]) will be conducted at pre-specified time points. In the event of treatment discontinuation, participants will continue to be followed and will be encouraged, though not required, to complete any remaining study assessments to minimize the occurrence of missing data.

Days 4-5 (72-96 hours): Predischarge Period Participants will remain inpatient for approximately 24 hours after the last scheduled study drug administration. Participants will complete a Patient Global Assessment (PGA) of satisfaction with study treatment at 84 (±2) hours or early discontinuation. During this period, participants may be administered standard of care to manage their pain, which will be recorded as concomitant medications. Pain intensity, PK, and safety assessments will be conducted at pre-specified time points until discharge on Day 5 (~96 hours).

Outpatient and Follow-up Phases Before discharge from the study center, study personnel will dispense a prescription for pain medication (if necessary) and an outpatient participant diary. Participants will be instructed to record use of any concomitant medications and adverse events (AEs) experienced after discharge in their outpatient participant diaries. Participants will also record their worst pain intensity in the last 24 hours at the end of each day and their current ("right now") pain intensity prior to use of any medication taken for pain. Participants will be instructed to return the outpatient participant diaries to study personnel at the follow-up visit, scheduled to occur 7 to 9 days after the abdominoplasty procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must provide written informed consent prior to the initiation of any protocol specific procedures.
2. Male or female participant, between 18 and 75 years of age, inclusive, at the time of Screening.
3. Participant must be scheduled to undergo a full abdominoplasty procedure without liposuction with no collateral procedures.
4. Participant must have physical status rated as I-II on the American Society of Anesthesiologists rating scale.
5. Participant must have a body mass index (BMI) within 18.0 to 32.0 kg/m2, inclusive (minimum weight of at least 50.0 kg).
6. If female, participant must be either not of childbearing potential (defined as postmenopausal for at least 1 year and confirmed with follicle stimulating hormone [FSH] >40 mIU/mL as deemed necessary by the investigator, or surgically sterile [bilateral tubal ligation, bilateral oophorectomy, or hysterectomy]) or participant must use a medically acceptable method of birth control (oral or transdermal hormonal contraceptives; vaginal ring; contraceptive implant or injection; intrauterine contraceptive system [with or without hormone]; condom and spermicidal foam; heterosexual abstinence; or sterilization of partner) from 30 days prior to Screening through 90 days after the last study drug administration. Heterosexual abstinence is considered to be a highly effective method only if the participant agrees to refrain from heterosexual intercourse during the entire period from 30 days prior to Screening to 90 days after the last study drug administration.
7. If male, participant must agree to use medically acceptable methods of contraception (diaphragm/sponge/condom with spermicide, vasectomy); female sexual partners of childbearing potential must be using and willing to continue using medically acceptable contraception (i.e., oral or transdermal hormonal contraceptives, vaginal ring, contraceptive implant or injection intrauterine contraceptive system [with or without hormone]) from Screening and for at least 90 days after the last study drug administration.
8. Must be able to speak, read, and understand English or Spanish sufficiently to allow completion of all study assessments.
9. Participant must be willing and able to follow study instructions and be likely to complete all study requirements.

Exclusion Criteria:

1. Participant has a history or presence of a clinically significant abnormality, as assessed by physical examination, medical history, electrocardiograms (ECGs; including a median QT interval corrected for heart rate [Fridericia; QTcF interval] of >450 milliseconds if male or >470 milliseconds if female at Screening and pre-operatively based on triplicate ECG; a repeat triplicate test is permitted and the median QTcF value will be used to determine eligibility), vital signs, or laboratory values, which, in the opinion of the investigator, would jeopardize the safety of the participant or the validity of the study results. Laboratory tests may be repeated once (one time) at Screening only, after approval by the medical monitor, if the investigator determines that the abnormal laboratory finding(s) was erroneous or caused by a temporary medical condition, for example, an acute infection, or by the temporary use of a prior medication.
2. Participant has a significant cardiac (e.g., ischemia or infarct, complete bundle branch blocks, symptomatic arrhythmias or predominantly non-sinus-conducted rhythm), pulmonary, gastrointestinal, endocrine, metabolic (except diabetes mellitus [A1c ≤7.0]), neurological, or psychiatric disorder (resulting in disorientation, memory impairment or inability to report accurately; for instance, schizophrenia, Alzheimer's disease), or any other clinically significant disease that, in the investigator's opinion, may affect efficacy or safety assessments, or that may compromise participant safety during trial participation.
3. Participant has a history of malignancy within the past 2 years, with the exception of basal cell carcinoma that has been treated and is no longer present.
4. Participant has a history or presence of acute respiratory depression, moderate or severe chronic pulmonary disease, cor pulmonale, delirium tremens, central nervous system (CNS) depression, or increased cerebrospinal or intracranial pressure.
5. Participant has a documented history of, or currently active, seizure disorder (excluding febrile seizures in childhood), or history of clinically significant head injury or syncope of unknown origin.
6. Participant has a current painful condition that could confound the interpretation of efficacy, safety, or tolerability data in the study, in the opinion of the investigator.
7. Participant has a history or presence of obstructive sleep apnea.
8. Participant has a known history of or presence of trypsin deficiency.
9. Participant has a history of acute or severe bronchial asthma, hypercarbia, or hypoxia.
10. Participant has any chronic gastrointestinal disease or major previous abdominal surgery (e.g., previous abdominoplasty surgery, Billroth procedure, enteroanastomosis, or bariatric surgery, including gastric bands and gastric sleeves, gastric bypass) that might affect the absorption, distribution, metabolism, or excretion of PF614. Prior cholecystectomy is allowed if the procedure was >1 year prior to Screening. Prior Caesarean section is allowed if the participant does not have altered sensation to the scar area.
11. Participant has a history of pancreatitis, pancreatic insufficiency, gastric ulcers, or gastrointestinal bleeding.
12. Participant has evidence of clinically significant hepatic or renal impairment, including alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3× the upper limit of normal (ULN), bilirubin >2× ULN, estimated creatinine clearance <60 mL/min (estimated by the 2021 Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] creatinine equation).
13. Participant has used chronic opioid therapy, defined as >15 mg oral morphine equivalent units per day, for >3 out of 7 days per week, for >1 month, within 12 months prior to first study drug administration.
14. Participant has used any analgesic medication within 5 half-lives (or, if half-life is unknown, within 48 hours) before the abdominoplasty procedure, or has used chronic non-steroidal anti-inflammatory drug (NSAID) therapy, defined as daily use for >2 weeks within 2 months prior to first study drug administration (aspirin ≤325 mg daily is permitted for cardiovascular prophylaxis if the participant has been on a stable regimen for ≥30 days before the abdominoplasty procedure).
15. Participant has used systemic steroid therapy within 3 months prior to first study drug administration, excluding over-the-counter (OTC) corticosteroid nasal spray products.
16. Participant has used any enzyme-modifying drugs or products, including strong inhibitors of cytochrome P450 (CYP) 3A4 and 2D6 enzymes (e.g., clarithromycin, itraconazole, ketoconazole, nefazodone, posaconazole, telithromycin, voriconazole, cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, diltiazem, and human immunodeficiency virus [HIV] antivirals) or strong inducers of CYP enzymes (e.g., rifampin, phenytoin, carbamazepine, phenobarbital, and St. John's Wort) within 30 days of first study drug administration.
17. Participant has used medications that, in the opinion of the investigator, could affect the analgesic response (such as central alpha-adrenergic agents [clonidine and tizanidine], antiepileptic drugs, gabapentinoids, benzodiazepines, antidepressants, neuroleptic agents or other antipsychotic agents) that are not stably dosed within at least 30 days prior to first study drug administration. Antidepressants are permitted if prescribed for anxiety or depression and doses have been stable for at least 30 days.
18. Participant has used a glucagon-like peptide-1 (GLP-1) receptor agonist, such as semaglutide, within 30 days prior to first study drug administration.
19. Participant is unable to discontinue any of the prohibited medications (Section 9.7.1).
20. Participant has a history or presence of any substance or alcohol use disorder, as defined by the Diagnostic and Statistical Manual of Mental Disorders - 5th Edition, Text Revision (DSM V TR).
21. Participant has a positive urine drug screen (UDS) or alcohol breathalyzer test at Screening (other than THC) or on the day of the abdominoplasty procedure. A positive UDS resulting from use of a prescribed medication not prohibited by the protocol may be allowed if, in the opinion of the investigator, the medication will not interfere with the study.
22. Participant has a history of suicidal ideation or suicidal behavior in the past 12 months, as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS; baseline version).
23. Participant has a history of allergy or hypersensitivity to any opioid analgesics, anesthetics, ondansetron, acetaminophen, or NSAIDs.
24. Female participant is currently pregnant (positive pregnancy test) or lactating, or is planning to become pregnant within 30 days of last study drug administration.
25. Participant is positive for hepatitis B surface antigen (HBsAg), hepatitis C, or HIV.
26. Participant has previously participated in a clinical trial using PF614.
27. Participant has received any investigational drugs or devices within 4 weeks (or 5 times the half-life of the drug, if known) prior to first study drug administration.
28. Participant has any medical condition that, in the opinion of the investigator, might interfere with the study procedures or data integrity or compromise the safety of the participant. Medical records may be requested at the opinion of the Investigator.
29. Participant is an employee of the sponsor or research site personnel directly affiliated with this study, or is their immediate family member, defined as a spouse, parent, child or sibling, whether biological or legally adopted.
30. Participant who, in the opinion of the investigator, is considered unsuitable or unlikely to comply with the study protocol for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Pain NRS-R area under the curve through 48 hours (AUC4-48) | 4-48 hours
  Pain at rest

SECONDARY OUTCOMES:
Pain NRS-A area under the curve through 48 hours (AUC4-48) | 4-48 hours
  Pain with activity
Pain NRS-R and NRS-A | 4-96 hours
  Partial AUCs (AUC4-12, AUC4-24, AUC4-36, AUC4-72, AUC12-24, AUC24-36, AUC36-48, AUC24 48, AUC48-72, AUC72-84, AUC72-96); AUC4-84; AUC4-96
Time to first use of rescue opioid medication | 0-96 hours
  Time to first use of rescue opioid medication through 96 hours
Total rescue opioid consumption through 24, 48, and 72 hours | 72 hours
  Use of rescue opioid medication for up to 72 hours after surgery
Proportion of participants who take at least 1 dose of rescue opioid medication | Up to 12, 24, 36, 48, and 72 hours
  Need for opioid rescue medication
Total rescue opioid consumption 72 through 96 hours | 0-96 hours
  Need for rescue opioid medication
Proportion of participants who discontinue from the inpatient treatment period early for any reason | 5 days
  Discontinuations
Scores on PGA of satisfaction with study treatment | 96 hours
  Patient Global Assessment (PGA) of study treatment

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - CenExel / Atlanta Center for Medical Research (ACMR), Atlanta, Georgia
  - HD Research - Memorial Hermann Surgery Center, Houston, Texas
  - CenExel / JBR, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: (In preparation)

REFERENCES:
- [Background] Kirkpatrick DL, Schmidt WK, Morales R, Cremin J, Seroogy J, Husfeld C, Jenkins T. In vitro and in vivo assessment of the abuse potential of PF614, a novel BIO-MD prodrug of oxycodone. J Opioid Manag. 2017 Jan/Feb;13(1):39-49. doi: 10.5055/jom.2017.0366. PMID 28345745
- [Background] Kirkpatrick DL, Evans C, Pestano LA, Millard J, Johnston M, Mick E, Schmidt WK. Clinical evaluation of PF614, a novel TAAP prodrug of oxycodone, versus OxyContin in a multi-ascending dose study with a bioequivalence arm in healthy volunteers. Clin Transl Sci. 2024 Mar;17(3):e13765. doi: 10.1111/cts.13765. PMID 38511523
- See also: Ensysce Biosciences home page — https://ensysce.com/